CLINICAL TRIAL: NCT01526369
Title: A Phase III Randomized Study of TH (Paclitaxel and Trastuzumab) Versus THL (Paclitaxel, Trastuzumab and Lapatinib) in First Line Treatment of HER2-positive Metastatic Breast Cancer
Brief Title: A Randomized Study of TH Versus THL in First Line Treatment of HER2-positive Metastatic Breast Cancer
Acronym: TH V THL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 11-10
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2-positive metastatic breast cancer.
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel; Lapatinib

ARMS (2):
- Paclitaxel and Trastuzumab (Active Comparator): Weekly paclitaxel (80mg/m², for 3 weeks of a 4 week cycle) + trastuzumab (8mg/kg loading dose on cycle 1 day 1 and 4mg/kg every 2 weeks) until disease progression, unacceptable toxicity or consent withdrawal.
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel
- Paclitaxel, Trastuzumab and Lapatinib (Experimental): Weekly paclitaxel (80 mg/m², for 3 weeks of a 4 week cycle) + trastuzumab (8 mg/kg loading dose on cycle 1 day 1 and 4 mg/kg every 2 weeks)
  + lapatinib (1,000 mg daily), until disease progression, unacceptable toxicity or consent withdrawal.
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel; Drug: Lapatinib

INTERVENTIONS:
Drug: Trastuzumab
Drug: Paclitaxel
Drug: Lapatinib
  Arms: Paclitaxel, Trastuzumab and Lapatinib

SUMMARY:
The proposed phase III randomised trial will compare the efficacy of trastuzumab and paclitaxel with trastuzumab, paclitaxel and lapatinib in first line treatment of HER2 positive metastatic breast cancer. The investigators will also examine potential predictive biomarkers of response to trastuzumab and lapatinib in pre-treatment biopsy samples and serum samples.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedures
2. Female age 18 years or greater.
3. ECOG Performance Status of 0 or 1.
4. Histologically or cytologically-confirmed invasive metastatic breast cancer.
5. Patients must have measurable disease according to RECIST criteria Version 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral CT scan,MRI, or calipers by clinical exam.
6. Tumour shows HER2 over-expression (3+ by IHC and/or FISH + ) by testing of the primary tumour and if available the biopsied metastatic lesion
7. Patients who received prior radiotherapy must have completed it at least 4 weeks before registration and recovered from all treatment-related toxicities.
8. Cardiac ejection fraction within the institutional range of normal as measured by MUGA or ECHO within 14 days prior to registration. Note that baseline and on treatment scans should be performed using the same modality and preferably at the same institution.
9. Adequate haematological, hepatic, and renal function.

   * Haemoglobin ≥ 9g/dL
   * Neutrophils (ANC/AGC) ≥1500/mm³ (1.5 x 10^9/L)
   * Platelets ≥ (100 x 10^9/L)
   * Total bilirubin ≤ 1.5mg/dL (25.65 μmol/L)
   * Both ALT (SGPT) and AST (SGOT) ≤ 3 x ULN with or without liver Metastasis
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Serum creatinine ≤1.5 ULN or calculated creatinine clearance (CrCl) ≥ 30mL/min according to the Cockcroft and Gault formula (Appendix K)
10. Able to swallow and retain oral medication.
11. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. Female patients of childbearing potential must have pregnancy excluded by urine or serum beta-HCG testing within 7 days prior to registration.
12. Estimated life expectancy greater than 12 weeks

Exclusion Criteria:

1. Prior systemic therapy for metastatic disease (except one line of hormonal therapy for metastatic disease without trastuzumab).
2. Recurrence within 12 months from completion of adjuvant chemotherapy to the development of metastatic disease.
3. Recurrence within 6 months from completion of adjuvant trastuzumab to the development of metastatic disease.
4. Prior lapatinib treatment.
5. Peripheral neuropathy ≥ grade 2
6. Patients with known CNS metastasis should be excluded from this clinical trial
7. Prior radiotherapy to more than half of the bony pelvis.
8. Uncontrolled or symptomatic angina, uncontrolled arrhythmias, congestive heart failure, a documented MI within 6 months prior to registration or any other cardiac disorders, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient .
9. Immediate or delayed hypersensitivity or untoward reaction to paclitaxel, trastuzumab, or other related compounds, or to drugs chemically related to lapatinib (including other anilinoquinazolines, e.g. gefitinib (Iressa®) and erlotinib (Tarceva®), or other chemically-related compounds).
10. Pregnant or breastfeeding women are excluded from this study.
11. Patients should not be receiving any other investigational agents (within 30 days prior to registration) or receiving concurrent anticancer therapy.
12. Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors (Table 9).
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
14. Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
15. Have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
16. Concurrent treatment with ovarian hormone replacement therapy. Prior treatment must be stopped prior to registration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-02-13 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 9 months

SECONDARY OUTCOMES:
Overall Survival | 30 months

CONTACTS AND LOCATIONS:
Locations (35):
- Finland (2):
  - Helsinki University Hopsital, Helsinki
  - Kuopio University hospital, Kuopio
- CRLC Val d'Aurelle, Montpellier, France
- Interdisziplinäre Onkologische Zentrum München (IOZ München), Munich, Germany
- Ireland (10):
  - St Vincent's University Hospital, Dublin, Leinster
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St James's Hospital, Dublin
  - University Hospital Galway, Galway
  - Midwestern Regional Hospital, Limerick
  - Sligo General Hospital, Sligo
  - Waterford Regional Hospital, Waterford
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Oslo University Hopsital, Oslo, Norway
- Hospital Santa Maria, Lisbon, Portugal
- Spain (17):
  - Centro Oncologico de Galicia, A Coruña
  - Hospital Nuestra Senora de Sonsoles, Ávila
  - Hospital Infanta Cristina, Badajoz
  - Hospital Virgen de la Luz, Cuenca
  - Hospital General de Grannollers, Granollers
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Complejo Hospitalario Xeral Calde / Hospital Lucus Augusti, Lugo
  - H. Puerta de Hierro, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital de Mataro, Mataró
  - Hospital Infanta Cristina, Parla
  - Hospital Donostia, San Sebastián
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital General Universitario de Elche, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clinico Universitario 'Lozano Blesa', Zaragoza